CLINICAL TRIAL: NCT03721536
Title: Effects of Low-Flow Anesthesia on Hemodynamic Parameters and Oxygenation in Morbidly Obese Patients Undergoing Bariatric Surgery: A Prospective, Randomized Clinical Trial
Brief Title: Effects of Low-Flow Anesthesia on Hemodynamic Parameters and Oxygenation in Morbidly Obese Patients
Acronym: Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat AKBAS, Asst. Prof. Dr. Sedat Akbas, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: sedatakbas4
Record Dates: First submitted 2018-10-18; First posted 2018-10-26 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Morbid Obesity; Hemodynamic Instability; Bariatric Surgery Candidate
Keywords: Morbidly obese patients; Bariatric surgery; Arterial blood analysis
MeSH Terms: conditions — Obesity, Morbid | interventions — Heart Rate; Arterial Pressure; Oxygen Saturation; Blood Gas Analysis; Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-flow anesthesia (Active Comparator): Patients in low-flow anesthesia receive a fresh gas flow of 4 L/min for the first 10 minutes and were then maintain with a fresh gas flow of 0.75 L/min. Patients will be monitored for hemodynamic parameters during the perioperative period. Arterial blood gase will be analyzed for the oxygenation.
  Interventions: Diagnostic Test: hemodynamic parameters; Diagnostic Test: arterial blood gase
- normal-flow anesthesia (Active Comparator): Patients in normal-flow anesthesia received a fresh gas flow of 4 L/min for the first 10 minutes and were then maintained with a fresh gas flow of 1.5 L/min. Patients will be monitored for hemodynamic parameters during the perioperative period. Arterial blood gase will be analyzed for the oxygenation.
  Interventions: Diagnostic Test: hemodynamic parameters; Diagnostic Test: arterial blood gase

INTERVENTIONS:
Diagnostic Test: hemodynamic parameters — vital signs on the monitor including heart rate, mean arterial pressure, peripheral oxygen saturation and End-tidal Carbon Dioxide
  Other Names: heart rate; mean arterial pressure; peripheral oxygen saturation; End-tidal Carbon Dioxide
Diagnostic Test: arterial blood gase — Arterial blood gas including partial oxygen pressure and partial carbon dioxide pressure is an important routine investigation to monitor the acid-base balance of patients, effectiveness of gas exchange, and the state of their voluntary respiratory control.
  Other Names: partial oxygen pressure; partial carbon dioxide pressure

SUMMARY:
Low-flow anesthesia has been used for years with positive results, but its effects on hemodynamic parameters and oxygenation are not clearly known in high-risk morbidly obese patients who are prone to pulmonary dysfunction related to the obesity. Therefore, this prospective randomized study aimed to compare the effects of low-flow (0.75 L/min) and normal-flow (1.5 L/min) anesthesia on hemodynamic parameters and oxygenation in morbidly obese patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Low-flow anesthesia has several potential benefits. It improves the flow dynamics of the inhaled air, increase mucociliary clearance, maintain body temperature, reduce fluid loss, result in savings of up to 75% and reduce greenhouse gas emissions and reduce treatment costs (10 - 13). However, it is necessary to examine whether the reduction of fresh gas flow affects the quality and safety of anesthesia management, especially during high-risk operations such as laparoscopic bariatric surgery.

Low-flow anesthesia has been used for years with positive results, but its effects on hemodynamic parameters and oxygenation are not clearly known in high-risk morbidly obese patients who are prone to pulmonary dysfunction related to the obesity. Therefore, this prospective randomized study aimed to compare the effects of low-flow (0.75 L/min) and normal-flow (1.5 L/min) anesthesia on hemodynamic parameters and oxygenation in morbidly obese patients undergoing laparoscopic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients with American Society of Anesthesiology (ASA) scores of III-IV,
* Aged 18-65 years old,
* BMI>40

Exclusion Criteria:

* Pregnant
* Uncontrolled diabetes mellitus,
* Cardiovascular disease,
* Pulmonary disease,
* Cerebrovascular disease,
* Drug and alcohol addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The level of partial oxygen pressure | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  The level of partial oxygen pressure is measured as mmHg in arterial blood gase analysis

SECONDARY OUTCOMES:
Heart rate | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Heart rate is measured as beats/minute on the anesthesia monitor
Mean arterial pressure | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Mean arterial pressure is measured as mmHg on the anesthesia monitor
Peripheral oxygen saturation | From beginning of Anesthesia induction to the end of anesthesia (during perioperative period)
  Peripheral oxygen saturation is measured as percentage (%) on the anesthesia monitor

CONTACTS AND LOCATIONS:
Overall Officials: Sedat Akbas, Asst Prof, Study Director — Inonu University Medical Faculty
Locations (1):
- Sedat Akbas, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunn Geoffrey BA. Low-flow anaesthesia. Continuing Education in Anaesthesia Critical Care & Pain Volume 8, Issue 1, February 2008, Pages 1-4
- See also: Low-flow anaesthesia — https://doi.org/10.1093/bjaceaccp/mkm052

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT03721536/Prot_SAP_000.pdf